CLINICAL TRIAL: NCT07113769
Title: Explore Plasma Biomarkers and Platelet Morphological Signatures for Predicting Prognosis in Patients With Extracorporeal CardioPulmonary Resuscitation (ECPR) Using Multi-omics and Platelet Morphology Analysis
Brief Title: Plasma Biomarkers and Platelet Morphology of Extracorporeal CardioPulmonary Resuscitation
Acronym: ECPR
Status: Not yet recruiting | Type: Observational
Sponsor: Central China Fuwai Hospital of Zhengzhou University (Other)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Henan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Jianchao, Li, Principal Investigator, Central China Fuwai Hospital of Zhengzhou University
Other Study IDs: ljc2025 No.12
Record Dates: First submitted 2025-06-18; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-06

CONDITIONS: ExtraCorporeal Membrane Oxygenation (ECMO); Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — Plasma 、platelet
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CA patients who have fully recovered after receiving ECPR treatment
- CA patients with organ dysfunction after receiving ECPR treatment
- CA patients who died or suffered brain death after receiving ECPR treatment

SUMMARY:
Extracorporeal cardiopulmonary resuscitation (ECPR) constitutes a pivotal emergency intervention for cardiac arrest (CA) patients. However, current eligibility criteria and prognostic assessment metrics remain substantially limited, relying predominantly on clinical symptoms and physical signs while lacking objective biomarker data. Integrating reproducible, highly sensitive, and specific proteinaceous and metabolic indicators with ultrastructural platelet alterations may hold significant implications for both ECPR administration and prognostication in CA. Therefore, the purpose of this study is to identify the plasma proteomic and metabolomic characteristics of patients with refractory cardiac arrest before and after ECPR treatment, as well as the characteristics of platelet morphological and structural changes, to search for potential specific markers that can predict CA patients who may benefit from ECPR so as to optimize treatment selection.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70 years old (the age limit can be relaxed if the patient has good organ function and a good neurological prognosis after evaluation).
2. The cardiac arrest is witnessed, and bystanders perform traditional cardiopulmonary resuscitation (CPR), and the time interval from the occurrence of cardiac arrest to the start of traditional CPR is no more than 5 minutes.
3. The causes of cardiac arrest are reversible, such as cardiogenic, pulmonary embolism, severe hypothermia, drug poisoning, trauma, acute respiratory distress syndrome, etc.
4. After 20 minutes of traditional CPR, there is no restoration of spontaneous circulation or hemodynamic instability, or the restoration of spontaneous circulation occurs, but the spontaneous heart rhythm cannot be maintained.
5. The informed consent has been signed.

Exclusion Criteria:

1. Infectious diseases, such as hepatitis B, hepatitis C, AIDS, syphilis, etc.
2. Hematological diseases, such as hematological malignancies, aplastic anemia, idiopathic thrombocytopenic purpura (ITP), etc.
3. Malignant tumors in other systems except the hematological system.
4. Patients who have received massive plasma or platelet transfusions during hospitalization or recently.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients receiving ECPR will be included. The decision to perform an ECPR is made by the local protocol and clinical judgment of the attending physician.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
30 day mortality | Within 30 days after ECPR
Hospital survival | Within 30 days after ECPR

SECONDARY OUTCOMES:
Cerebral Performance Category (CPC) scale | 30 days after ECPR
Left Ventricular Ejection Fraction (LVEF) | Within 30 days after ECPR
PaO2/FiO2 ratio | Within 30 days after ECPR
Serum Bilirubin level | Within 30 days after ECPR
Creatinine | Within 30 days after ECPR

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Central China Cardiovascular Hospital, Zhengzhou, Henan, China